CLINICAL TRIAL: NCT06722495
Title: Efficacy and Safety of a Third-Course of Neoadjuvant Immunochemotherapy Combined With SBRT in Locally Advanced Head and Neck Squamous Cell Carcinoma Patients With Stable Disease After Two Treatment Courses: A Single-Arm Exploratory Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-804-02
Record Dates: First submitted 2024-11-06; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: SBRT; Neoadjuvant Immunochemotherapy; LA HNSCC

STUDY DESIGN:
Intervention Model Description: This is a single-arm exploratory clinical study aimed at evaluating the efficacy and safety of combining stereotactic body radiation therapy (SBRT) with subsequent treatments in patients with locally advanced head and neck squamous cell carcinoma (LA HNSCC) who are unresponsive to neoadjuvant immunochemotherapy. The study plans to enroll 20 patients diagnosed with stage III-IVb (AJCC 8th) LA HNSCC who have received two cycles of platinum-based chemotherapy and PD-1 inhibitor immunotherapy, but achieved stable disease (SD) according to RECIST 1.1 criteria. These patients will receive SBRT (8Gy*3F) during the third cycle of immunochemotherapy, followed by standard surgery and postoperative radiotherapy/chemoradiotherapy. The primary endpoint is the objective response rate (ORR) of the primary lesion after the third cycle, with secondary endpoints including overall ORR, pathologic complete response (pCR), major pathologic response (mPR), and partial pathologic response (pPR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3-Course of Neoadjuvant Immunochemotherapy combined with SBRT in LA-HNSCC with SD after 2-courses (Experimental): Stereotactic body radiation therapy added between 2-course and 3-course treatment.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patient will receive SBRT (8Gy*3F) in combination with the original regimen of neoadjuvant immunochemotherapy in course 3. Gross tumor target volume (GTV) based on the primary foci clearly identified by clinical and imaging examinations. The GTV was discharged 3 mm to generate a Planning target volume (PTV). the target area (PTV) was dosed accordingly to the PTV.

SUMMARY:
Neoadjuvant immunotherapy before surgery has shown good efficacy and safety in locally advanced HNSCC, particularly with the use of PD-1 inhibitors combined with chemotherapy, where some patients have achieved a high rate of pathological complete response. However, approximately 40% of patients respond poorly to neoadjuvant immunochemotherapy, with prolonged treatment courses failing to significantly improve outcomes, and some patients may even experience disease progression. For these patients, timely surgery or definitive radiotherapy combined with other well-tolerated therapeutic approaches is needed to improve pathological response rates, enhance long-term survival, and preserve organ function.

DETAILED DESCRIPTION:
In recent years, the introduction of PD-1 inhibitors has revolutionized cancer treatment, including head and neck squamous cell carcinoma (HNSCC). Data from The Cancer Genome Atlas (TCGA) shows HNSCC is one of the most immunogenic cancers, linked to immune dysfunction such as impaired immune cell function and antigen presentation defects. Immunotherapy, alone or combined with chemotherapy, has become the standard first-line treatment for recurrent or metastatic HNSCC, as supported by clinical trials like Keynote-040, Keynote-048, and CheckMate 141, which demonstrated improved patient outcomes.

There is also growing interest in neoadjuvant immunotherapy for locally advanced HNSCC. A phase II clinical trial (NCT03174275) showed that neoadjuvant camrelizumab combined with cisplatin and paclitaxel achieved a pathologic complete response (pCR) rate of 37% and a major pathological response (MPR) rate of 74%. Another trial combining PD-1 inhibitor tislelizumab with nab-paclitaxel, platinum, and fluorouracil reported an objective response rate (ORR) of 85.7% and a pCR rate of 42.9%.

In a retrospective analysis of 110 locally advanced oral cavity squamous cell carcinoma (OCSCC) patients treated at our institution, the ORR after two cycles of neoadjuvant immunochemotherapy was 55.4%, with 41% of patients showing stable disease (SD). Further treatment cycles did not improve outcomes for these patients, highlighting the need for alternative treatments for those unresponsive to neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years on the date of signing the informed consent form, male or female.
2. Histologically and imaging-confirmed T3-4a or N+M0 stage III-IVb (AJCC 8th) HNSCC, patients have received 2-courses of platinum-based chemotherapy and tirilizumab immunotherapy, and whose efficacy is assessed as Stable Disease (SD).
3. Life expectancy is at least 3 months.
4. ECOG PS 0-1。
5. Haematological analysis： 5.1 Absolute neutrophil count (ANC) ≥1.5×10^9/L without granulocyte colony-stimulating factor in the last 14 days； 5.2 Absolute T-lymphocyte value ≥ 0.5 times the lower limit of normal value； 5.3 Platelets ≥100×10^9/L without transfusion or platelet-boosting drugs in the last 14 days； 5.4 Haemoglobin ≥90g/L without transfusion or erythropoietin use in the last 14 days.
6. Renal function:

   6.1 Creatinine clearance* (Ccr) ≥60 mL/min; *Ccr will be calculated using the Cockcroft-Gault formula: Ccr = (140-age) × body weight (kg) / [0.818 (0.85 for males, 0.85 for females) × blood creatinine (SCr, umol/L) ] or Ccr = (140-age) × body weight (kg)/ [72 × blood creatinine (SCr, mg/dL) ]; 6.2 Creatinine ≤ 1.5 × upper limit of normal (ULN)； 6.3 Routine urinalysis suggests urinary protein ≤ +; 6.4 Quantitative 24-hour urine protein <1.0g.
7. Liver function:

   7.1 Serum total bilirubin (TBil) ≤ 1.5 × ULN; 7.2 AST and ALT ≤ 2.5 × ULN, ≤ 5 × ULN for liver metastases, and TBil ≤ 3 × ULN.
8. Coagulation: international normalised ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
9. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects may be enrolled if total T3 (or FT3) and FT4 are within the normal range.
10. Cardiac enzyme profiles within the normal range (enrolment is also permitted if the investigator's combined judgement is that it is a purely laboratory abnormality of no clinical significance).
11. Patients must be able to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Hypersensitivity to any of the antineoplastic therapeutic drug components of this research.
2. Those who have previously suffered from other malignant tumours and have received radiotherapy.
3. have uncontrolled clinical symptoms or cardiac disease including, but not limited to, symptomatic congestive heart failure (Grade 2 and above as determined by the New York Heart Association's Functional Class), unstable angina pectoris, acute myocardial ischaemia, and poorly controlled cardiac arrhythmias. Past history of myocarditis and cardiomyopathy.
4. Active autoimmune disease requiring systemic therapy (e.g., use of disease-mitigating drugs, glucocorticoids, or immunosuppressants). Alternative therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy.
5. History of (non-infectious) pneumonia requiring steroids or current pneumonia.
6. Have active tuberculosis.
7. History of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to first dose or current clinically active interstitial lung disease.
8. Active or uncontrolled infection requiring systemic therapy.
9. History of human immunodeficiency virus (HIV) infection (e.g., HIV-positive).
10. Liver disease such as cirrhosis, decompensated liver disease; known active hepatitis B (e.g., hepatitis B surface antigen (HBsAg) positive and HBV-DNA > upper limit of normal in the laboratory of the research centre) or active hepatitis C virus infection (e.g., HCV antibody positive and HCV RNA level above the lower limit of detection).

    *Note: Hepatitis B subjects meeting the following criteria may also be enrolled: 10.1 HBV viral load <1000 copies/ml (200 IU/ml) prior to the first dose, and subjects should receive anti-HBV therapy throughout the study treatment period to avoid viral reactivation; 10.2 In subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is needed.
11. Have an active bleeding disorder or other history of severe bleeding.
12. Allogeneic organ transplantation (except corneal transplantation) or allogeneic haematopoietic stem cell transplantation.
13. Pregnant or breastfeeding, or preparing to become pregnant during the trial period.
14. Medical, psychological, or social condition that may interfere with the subject's participation in the research or affect the assessment of the results; or other conditions that, in the opinion of the investigator, make enrolment inappropriate, or that, in the opinion of the investigator, present other potential risks that make participation in this research inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-24 (Estimated); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 weeks after the 3rd course of Neoadjuvant immunochemotherapy + SBRT, including by imaging assessment.
  Proportion of subjects containing complete response and partial response, i.e., the sum of the diameters of the target lesions is at least 30% smaller compared to baseline, derived from the RECIST v1.1 criteria at 3 weeks after the 3rd course of Neoadjuvant immunochemotherapy + SBRT, including by imaging assessment.

SECONDARY OUTCOMES:
Overall response rate | 3 weeks after the 3rd course of Neoadjuvant immunochemotherapy + SBRT, including by imaging assessment.
  The percentage of patients with a best overall response of CR or PR relative to the efficacy evaluable population.
Pathological complete response | 10days after surgery
  No surviving tumor cells are found in a sample of a completely resected tumor.
Major pathologic response | 10days after surgery
  Percentage of residual viable tumor cells ≤10% in samples of completely resected tumors.
Pathological partial response | 10days after surgery
  Percentage of residual viable tumor cells >10%, ≤70% in samples of completely resected tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No